CLINICAL TRIAL: NCT04143087
Title: A Multicenter, Open-access Study of CML-CP Patients Treated With Effective TKIs at Least 5 Years and MR4.5(BCR/ABLIS<0.0032%) Maintenance More Than 18 Months Who Treatment With Half TKIs or Discontinue
Brief Title: Withdrawal or Reduction TKIs in CML-CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xuna, Associate chief physician, Nanfang Hospital, Southern Medical University
Other Study IDs: TKIs-cml-002
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: MMR on 12 Month

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Withdrawal TKIs
  Interventions: Drug: withdrawal TKIs or halve TKIs
- halve TKIs
  Interventions: Drug: withdrawal TKIs or halve TKIs

INTERVENTIONS:
Drug: withdrawal TKIs or halve TKIs — Stop TKIs or treated by half TKIs

SUMMARY:
Compare MMR on 12 month treated with half TKIs(including imatinib, dasatinib, and nilotinib) or TKIs withdrawal.

DETAILED DESCRIPTION:
1. Chronic myeloid leukemia-Chronic phase(CML-CP) patients treated with receive effective Tyrosine kinase inhibitor -TKI(including imatinib, dasatinib and nilotinib) for more than 5 years, and patients with BCR/ABLIS continuous negative in the last 18 months were randomly admitted to maintain the original effective TKI by half or stop taking .
2. Q-pcr detected BCR/ABLIS in peripheral blood once every month, once every two months after half a year, and continuously monitored for 12 months.
3. If the patients detected molecular recurrence (loss of MMR, BCR/ABLIS > 0.1%), the original dose of TKI should be administered again.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, gender is not limited;
2. Diagnosed CML chronic phase and effective TKI(including imatinib, dasatinib, and nilotinib) was continued for more than 5 years
3. Q-PCR monitored BCR/ABLIS duration < 0.0032% in the last 18 months
4. Informed consent of the patient or his legal representative

Exclusion Criteria:

1. Patients had history of CML-AP or CML-BC
2. CML patients with previous or current ABL kinase mutations
3. CML Patients who have received allogeneic hematopoietic stem cell transplantation
4. CML Patients who have received immunotherapy (except interferon, including car-t and other cellular immunotherapy)
5. Woman who is pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed CML chronic phase,Age 18-70 years old,gender is not limited
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
MMR(BCR/ABL IS<0.01) on 12 moth | 12 moth
  Half dose TKIs or discontinue TKIs treatment

CONTACTS AND LOCATIONS:
Locations (1):
- NanfangH, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Luo J, Du X, Lou J, Wu J, Ma L, Huang J, Wang L, Tu C, Liu Z, Chen L, Tan Y, Luo D, Liang H, Yin C, Cao R, Zhou X, Liu Q, Liu X, Xu N. De-escalation or discontinuation of tyrosine kinase inhibitor in patients with chronic myeloid leukemia: A multicentral, open-label, prospective trial in China. EJHaem. 2022 Sep 19;3(4):1220-1230. doi: 10.1002/jha2.550. eCollection 2022 Nov. PMID 36467815